CLINICAL TRIAL: NCT03128762
Title: Circulating Innate Lymphoid Cell Type 2 (ILC2) Levels and Asthma: a Case-control Study
Acronym: ILC2-Asthma
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9243; 2013-A01443-42 (Other: RCB number)
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients in this group are asthmatic (see inclusion/exclusion) criteria.
  Intervention: ILC2 levels in blood
  Interventions: Biological: ILC2 levels in blood
- Controls: Controls are non-asthmatic subjects that are age and gender matched to asthma cases.
  Intervention: ILC2 levels in blood
  Interventions: Biological: ILC2 levels in blood

INTERVENTIONS:
Biological: ILC2 levels in blood — The levels of circulating ILC2 cells relative to other lymphocytes will be determined via flow cytometry

SUMMARY:
The primary objective of this study is to demonstrate differences in ILC2 blood levels between asthma patients and control patients.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

To show that ILC2 levels differ between asthma patients with a "TH2" (helper T cell type 2) profile and asthma patients with a "non-TH2" profile. A TH2 profile is defined as (for a given patient):

* circulating eosinophils > 500 mm^3 at least once during the year AND
* positive allergy skin or specific IgE (Immunoglobulin E) test AND
* induced sputum eosinophil level >3% of leukocytes AND
* exhaled nitric oxide > 25 ppb.

To study the variation in ILC2 levels over time among asthma patients who obtained a good level of control compared to other patients. A good level of control is defined as:

* no exacerbations during 6 months of followup (an exacerbation is defined as the un-planned need for care that modifies the patient's prescription for >48h)
* FEV1 (forced expiratory volume in 1 second) value current / FEV1 best value > 0.8
* symptom levels correspond to an ACQ (Asthma Control Questionnaire) questionnaire score of < 0.75 over the last 7 days

ELIGIBILITY:
Inclusion Criteria for Cases:

* The subject has given his/her informed consent and signed the consent form
* The subject is affiliated with or beneficiary of a medical insurance system
* The subject has had asthma for over a year
* The following are present in the patient's medical file: (i) a positive methacholine test (PC20 < 16 mg/ml) OR (ii) reversibility > 200 ml and 12% of the FEV1 after inhaling 400 µg or less of a short acting bronchodilator.
* Treatment with >= 1000 µg inhaled beclometasone equivalents

Exclusion Criteria for Cases:

* The subject is pregnant
* The subject is breastfeeding
* The subject is participating in another interventional study
* The subject has participated in another study in the 3 months preceding inclusion
* The subject is in an exclusion period determined by a previous study
* The subject is under judicial protection or is an adult under any kind of guardianship
* The subject refuses to sign the consent
* It is impossible to correctly inform the subject
* The subject cannot fluently read French
* Chronic respiratory disease present, known or suspected (other than asthma)
* Treated with Montelukast

Inclusion Criteria for Controls:

* The subject has given his/her informed consent and signed the consent form
* The subject is affiliated with or beneficiary of a medical insurance system

Exclusion Criteria for Controls:

* The subject is pregnant
* The subject is breastfeeding
* The subject is participating in another interventional study
* The subject has participated in another study in the 3 months preceding inclusion
* The subject is in an exclusion period determined by a previous study
* The subject is under judicial protection or is an adult under any kind of guardianship
* The subject refuses to sign the consent
* It is impossible to correctly inform the subject
* The subject cannot fluently read French
* Any kind of bronchial problem
* Smokers
* Chronic respiratory disease present, known or suspected
* Treated with Montelukast

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This case-control study compares cases (asthma patients) with healthy control subjects. Patients and controls are matched by sex and age (+- 5 years).
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-06-25 (Actual); Primary Completion 2015-04-14 (Actual); Study Completion 2015-06-23 (Actual)

PRIMARY OUTCOMES:
% ILC2 cells among total blood lymphocytes | Day 0
  Determined by flow cytometry

SECONDARY OUTCOMES:
% ILC2 cells among total blood lymphocytes | 6 months
  Determined by flow cytometry; Asthma patients only.